CLINICAL TRIAL: NCT01262495
Title: Testicular Tissue Viability After Cryopreservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: hadassah, hadassah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: kabiri HMO-CTIL
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Fertility
MeSH Terms: interventions — Cryopreservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- orchidectomy (Other): as specified in the summary
  Interventions: Other: cryopreservation

INTERVENTIONS:
Other: cryopreservation — cryopreservation of testicular tissue

SUMMARY:
we will use testicular tissue from patient who underwent orchidectomy due to medical reasons and test the viability of the tissue after cryopreservation and de-freezing.

ELIGIBILITY:
Inclusion Criteria: male patient undergo orchidectomy -

Exclusion Criteria: non viable testicular tissue

-

Ages: 15 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
viable tissue after cryopreservation | 1/1/2011 - 30/12/2012

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel